CLINICAL TRIAL: NCT00333190
Title: CD8+ T Cell Depletion as Graft Versus Host Disease Prophylaxis After HLA-Matched Unrelated Donor Non-myeloablative Peripheral Blood Stem Cell Transplantation
Brief Title: CD8+ T Cell Depletion for GVHD Prophylaxis After Peripheral Blood Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Vincent T. Ho, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-151
Record Dates: First submitted 2006-05-25; First posted 2006-06-02 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Hematologic Malignancy; AML; ALL; CML; Multiple Myeloma; NHL; Hodgkin's Lymphoma
Keywords: stem cell transplant; graft versus host disease; GVHD; CD+8 T cell depletion
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Hodgkin Disease; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CD+8 T cell depletion — CD8 depleted product Given through central line after treatment with fludarabine and busulfex intravenously for 4 days

SUMMARY:
The purpose of this trial is to determine if selectively removing only a small subset of T cells, called CD8+ T cells, is safe and if it can reduce the risk of graft versus host disease (GVHD) without losing the anti-cancer effects.

DETAILED DESCRIPTION:
* The patient will be admitted to the hospital once a good donor is found for chemotherapy and stem cell transplant. The patient will remain in the hospital for 8 days and will receive two chemotherapy drugs (fludarabine and Busulfex) intravenously once each day for 4 days.
* On the third day after the patient has finished chemotherapy, the donor cells should arrive at Dana-Farber Cancer Institute and the lab will remove CD8 cells. Then the product will be given to the patient through a central line. If there are not enough stem cells in the donor product, then the CD8 cells will not be taken out, and the patient will get the whole product.
* Just before and after the transplant, the patient will also take tacrolimus and methotrexate to help prevent GVHD. Tacrolimus is a pill that will be taken orally two times a day. Methotrexate is a chemotherapy drug that is given intravenously on days 1, 3 and 6 after the transplant. In addition to the these drugs, participants will also take antibiotics to prevent infection and Filgrastim (G-CSF, neupogen) until their white blood cell counts are better.
* After the stem cell infusion, check-ups and blood tests will be performed at least once a week for 1 month. At about one month, a bone marrow biopsy to look for the donor's cells in the participants bone marrow will be performed. After the 1-month evaluation, the patient will be seen at least every 2 weeks with another bone marrow biopsy at 3-4 months after the transplant.
* After the patient is past 100 days since transplant, they will be followed in the clinic and have blood work done at least once a month until 6 months post transplant.
* The trial will end at 6 months after the transplant, but patients will be tracked for the rest of their life to look at long-term effects of this transplant.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic malignancies that are candidates for allogeneic non-myeloablative stem cell transplantation
* AML or ALL in first or subsequent remission, or in resistant or untreated relapse with marrow blast < 20% of cellularity
* CML in first or subsequent chronic phase, or accelerated phase
* Myelodysplastic syndrome with < 20% marrow blasts
* NHL or Hodgkin's lymphoma in second or greater remission, or partial remission after salvage therapy, and in patients with marrow involvement, <20% involvement in BM
* CLL RAI stage 2-4, which has progressed after initial fludarabine containing therapy, and BM involvement of < 20%
* Multiple myeloma stage II-III, in first or subsequent plateau phase with <20% BM plasma cells
* Available unrelated donor who is fully HLA matched at HLA-A,B,C and DRB1
* Age 18 or greater
* Performance status 0-2
* Life expectancy of > 100 days
* No HLA-matched related donor available

Exclusion Criteria:

* Myeloproliferative disorders other than CML
* MDS with myeloproliferative features, or CMML
* High grade Burkitts or Burkitts-like Non-Hodgkin's lymphoma
* Prior allogeneic stem cell transplant
* Active CNS involvement with disease
* Uncontrolled infection
* Pregnancy
* Evidence of HIV infection
* Heart failure uncontrolled my medications
* Total bilirubin > 2.0 mg/dl that is due to hepatocellular dysfunction
* AST > 2 x institutional upper limit of normal
* Serum creatinine > 2.0 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the initial engraftment of HLA matched unrelated donor mobilized peripheral blood stem cells depleted of CD+8 cells. | 2 years

SECONDARY OUTCOMES:
To assess sustained engraftment | 2 years
to determine the incidence of GVHD | 2 years
to assess disease relapse. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent T. Ho, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts